CLINICAL TRIAL: NCT07309770
Title: Trastuzumab Rezetecan in Advanced Solid Tumors Refractory to Standard Therapies: A Multicenter, Single-Arm, Phase II Study With Multiple Cohorts
Brief Title: Trastuzumab Rezetecan in Advanced Solid Tumors Refractory to Standard Therapies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Sheng Zhang, Prof., Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1811-US-03
Record Dates: First submitted 2025-09-28; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: Urachal Cancer; Advanced Solid Tumor Cancer; Antibody-drug Conjugates
Keywords: Antibody-Drug Conjugates; Rare tumor; Extra-mammary Paget disease; Urachal cancer; Trastuzumab Rezetecan
MeSH Terms: conditions — Urachal cancer; Paget Disease, Extramammary

STUDY DESIGN:
Intervention Model Description: single-group study,three cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group 1 (Experimental): Cohort1:Patients with histologically confirmed extramammary Paget's disease (EMPD) demonstrating HER2 expression (IHC ≥ 1+) and having unresectable locally advanced or metastatic disease.
  Cohort2: Patients with histologically confirmed locally advanced or metastatic rare solid tumors (such as sarcoma, urachal carcinoma, etc.) demonstrating HER2 expression (IHC ≥ 1+) , who have experienced disease progression on or after standard therapy, or for whom no standard therapy is available, and with at least one measurable lesion.
  Cohort3:Patients with histologically confirmed locally advanced or metastatic urothelial carcinoma demonstrating HER2 expression (IHC ≥ 1+) , who have experienced disease progression following first-line treatment with a PD-1/PD-L1 inhibitor in combination with Enfortumab Vedotin or Disitamab vedotin
  Interventions: Drug: SHR-A1811; Drug: Trastuzumab Rezetecan

INTERVENTIONS:
Drug: SHR-A1811 — Trastuzumab Rezetecan (SHR-A1811) is administered at a dose of 4.8 mg/kg every 21 days (q3w), constituting one treatment cycle.
Drug: Trastuzumab Rezetecan — Patients who have failed standard therapy are treated with Trastuzumab Rezetecan

SUMMARY:
This study is a single-center, multi-cohort, phase II clinical trial. Eligible patients with HER2-positive advanced solid tumors were enrolled after providing informed consent. A total of 90 patients were allocated into three cohorts (30 patients each): those with Extramammary Paget's Disease (EMPD), rare solid tumors, or urothelial carcinoma, who had experienced failure of standard treatment or for whom no standard treatment was available. The participant recruitment period was 12 months, and the follow-up duration was 12 months. All patients received Trastuzumab Rezetecan (SHR-A1811) at a dose of 4.8 mg/kg administered every three weeks (q3w). They were followed until disease progression, withdrawal from the study, loss to follow-up, or death, whichever occurred first. Tumor response was assessed radiologically every 6 weeks during treatment. Safety follow-up was conducted 30 days after the last dose, followed by survival follow-up every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign a written informed consent form.

Age ≥ 18 years.

Diagnosed with the corresponding advanced tumor confirmed by histology and/or cytology, combined with imaging or ultrasound assessment, and pathologically confirmed as HER2-positive (i.e., HER2 ≥ 1+ by immunohistochemistry [IHC]).

Cohort 1 only: Histologically confirmed extramammary Paget's disease (EMPD) with unresectable locally advanced or metastatic disease.

Cohort 2 only: Histologically confirmed locally advanced or metastatic rare solid tumor (e.g., sarcoma, urachal cancer) refractory to standard treatment or for whom no standard treatment is available.

Cohort 3 only: Histologically confirmed locally advanced or metastatic urothelial carcinoma with disease progression following first-line treatment with a PD-1/PD-L1 inhibitor combined with enfortumab vedotin or disitamab vedotin.

ECOG Performance Status: 0 to 2.

At least one measurable lesion (according to RECIST v1.1 criteria: non-nodal lesions with longest diameter ≥10 mm on CT scan, nodal lesions with short axis ≥15 mm on CT scan).

Hematological function:

Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L

Platelet count (PLT) ≥ 70 × 10⁹/L

Hemoglobin (HGB) ≥ 80 g/L

Hepatic function:

Serum total bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal (ULN)

Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × ULN (≤ 5 × ULN if liver metastases are present)

Serum albumin ≥ 28 g/L

Renal function:

Serum creatinine (Cr) ≤ 1.5 × ULN or Creatinine clearance ≥ 50 mL/min (calculated using the standard Cockcroft-Gault formula)

Coagulation function:

International Normalized Ratio (INR) ≤ 1.5 and/or Prothrombin Time (PT) ≤ 1.5 × ULN

Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN

Estimated life expectancy ≥ 3 months.

Use of medically approved contraception during the treatment period and for at least 120 days after the end of the study; sperm donation or cryopreservation for fertilization purposes is not allowed during this period.

Ability to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in this study:

Presence of any severe and/or uncontrolled disease, including:

Poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L).

≥ Grade 2 myocardial ischemia, myocardial infarction, arrhythmia (QTcF ≥ 470 ms), or ≥ Grade 2 congestive heart failure (New York Heart Association [NYHA] classification).

Active or uncontrolled severe infection (≥ CTCAE Grade 2 infection) requiring systemic antibacterial, antifungal, or antiviral treatment, including tuberculosis infection.

History of active tuberculosis.

Uncontrolled ascites, pericardial effusion, or pleural effusion requiring repeated drainage.

Active hepatitis (liver enzyme levels not meeting inclusion criteria; for Hepatitis B: HBV DNA ≥ 2000 IU/ml or ≥ 10⁴ copies/ml; for Hepatitis C: HCV RNA ≥ 2000 IU/ml or ≥ 10⁴ copies/ml; carriers with chronic hepatitis B virus [HBV DNA < 10⁴ IU/ml] may be enrolled if they receive concomitant antiviral therapy during the trial).

History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases.

Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

Known presence of brain metastases, leptomeningeal metastasis, spinal cord compression, or spinal metastasis.

Within 6 months prior to the first dose: history of esophageal/gastric varices, severe ulcer, unhealed wound, gastrointestinal perforation, abdominal fistula, intestinal obstruction, intra-abdominal abscess, acute gastrointestinal bleeding; extensive intestinal resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.

Presence of non-healing or poorly healed wounds, active ulcers.

Toxicity from previous antineoplastic therapy that has not resolved to ≤ Grade 1 per NCI CTCAE v5.0 (except for alopecia).

Major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or presence of long-term unhealed wounds or fractures.

History of severe hypersensitivity reaction to monoclonal antibodies; known allergy to the active components or excipients of the study drug(s).

Participation in another clinical trial within 4 weeks prior to the start of the study.

Administration of a live vaccine within 30 days prior to the first dose, or planned administration during the study.

History of severe allergy.

Bleeding tendency, coagulopathy, or undergoing thrombolytic therapy.

History of drug abuse or inability to discontinue use, or history of psychiatric disorders.

History of clear neurological or psychiatric disorders, such as dementia, epilepsy, or susceptibility to seizures.

Any condition that, in the investigator's judgment, seriously endangers subject safety, affects subject completion of the study (e.g., severe diabetes, thyroid disease, psychosis), may compromise subject safety or the ability to provide informed consent (including abnormal laboratory findings), or involves psychological, familial, sociological, or geographical conditions that may preclude compliance with the study protocol and follow-up plan.

Any other reason deemed by the investigator to make the subject unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2027-09-11 (Estimated); Study Completion 2028-03-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved CR or PR according to RECIST V.1.1 criteria. | Efficacy was assessed every 9 weeks for 1 year and every 12 weeks thereafter (assessed up to 3 years).
  Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Time from treatment start to progression by RECIST V.1.1. | From date of treatment until the date of first documented progression, assessed up to 100 months.
  Progression-free survival(PFS)
Time from treatment start to death of participants. | From date of treatment until the date of death from any cause, whichever came first, assessed up to 100 months.
  Overall Survival(OS)
Type, incidence, severity, onset and end time of adverse events (AE) evaluated according by the version 5.0 of NCI-CTCAE. | Began at 30 days (±7 days) after the last study treatment to 1 year.
  Evaluation of safety

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided